CLINICAL TRIAL: NCT01707641
Title: A Randomized Study on the Effects of Lactobacillus Brevis CD2 in the Prevention of Radio and Chemotherapy Induced Oral Mucositis in Head and Neck Cancer Patients.
Brief Title: Effect of Lactobacillus Brevis CD2 in Prevention of Radio-chemotherapy Induced Oral Mucositis in Head and Neck Cancer
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: S. Andrea Hospital (Other)
Responsible Party: Principal Investigator, Vitaliana De Sanctis, M.D. University Researcher, S. Andrea Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CD2 AIRO
Record Dates: First submitted 2012-10-12; First posted 2012-10-16 (Estimated); Last update posted 2014-05-20 (Estimated); Status verified 2014-05

CONDITIONS: Mucositis
MeSH Terms: conditions — Mucositis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- CD#2 (Active Comparator): patients will be asked to melt slowly in the mouth 6 lozenges per day, containing Lactobacillus brevis CD2
  Interventions: Dietary Supplement: CD#2
- bicarbonate sodium mouthwash (Active Comparator): patients will be asked to wash their mouth with bicarbonate several times per day
  Interventions: Other: bicarbonate sodium mouthwash

INTERVENTIONS:
Dietary Supplement: CD#2 — patient will be asked to take 6 lozenges every day and let it dissolve slowly in the mouth
  Other Names: Lozenge containing Lactobacillus brevis CD2
  Arms: CD#2
Other: bicarbonate sodium mouthwash — Patients will be asked to wash their mouth with bicarbonate sodium several times per day
  Arms: bicarbonate sodium mouthwash

SUMMARY:
Oral mucositis is a debilitating side effect for oncology patients and there is a clear need for new therapeutic options. The lozenges containing Lactobacillus brevis CD2 proved a potential new alternative for the prevention of grade III and IV mucositis. The main endpoint of this study is to verify if these lozenges taken 6 times a day may reduce the incidence of grade III and IV mucositis as well as increase the percentage of patients who will complete the radio-chemotherapy treatment.

DETAILED DESCRIPTION:
Mucositis is a debilitating side effect of radio and chemotherapy treatment in oncology patients. It is not only painful, but also can limit adequate nutritional intake and decrease the willingness of patients to continue the treatment. Furthermore, extensive mucositis may require additional nutritional supplementation, and narcotic analgesic increasing the cost of the therapy. Quality of life is impaired in patients who develop severe mucositis.

Clinically, it begins with asymptomatic redness and erythema and ultimately passing through different stages to large acutely painful contiguous pseudomembranous lesions with associated dysphagia and decreased oral intake. The common sites of oral mucositis are labial, buccal, soft palate, floor of mouth, and the ventral surface of the tongue. The loss of the epithelial cells exposes the underlying connective tissue with its associated innervations causing pain. Oral infections, which may be due to bacterial, fungal, or viruses may further exacerbate the mucositis as well as lead to systemic infections.

Treatment and prevention of therapy related mucositis is essential; unfortunately, the efficacy and safety of most of the regimen used have not been clearly established. Prophylactic measures employed are use of: chlorhexidine, saline rinses, soda bicarbonate rinses, acyclovir, and ice. For treatment of mucositis and its associated pain local anesthetic, diphenhydramine, nystatin, or sucralfate are used alone or in combination as mouthwash. Oral or parenteral narcotics are also used for pain relief.

There is a clear need for new therapeutic options for oral mucositis.

ELIGIBILITY:
Inclusion Criteria:

* male and female patients > 18 years of age
* Karnofsky Performance Status >70%
* pathological and histological diagnosis that confirms head and neck tumour
* patients eligible for radical radiotherapy and/or chemotherapy
* expected survival time > 6 months
* normal bone marrow function (neutrophil count >1500/cmm, platelet count > 100.000/CMM)
* serum creatine < 1.8mg/dl
* total bilirubin <2mg/dl
* GOT, GPT within 3 times the normal limit
* willingness to perform conventional 3D radiotherapy or intensive modulated radiation therapy with concurrent chemotherapy
* signed informed consent form

Exclusion Criteria:

1. Diagnosis of glottic tumour, parotid or salivary, larynx tumour.
2. Presence of metastasis, detected with contrast-enhances TC TB and/or PET/TC
3. Major surgery of the oral cavity within the last 4 weeks
4. Patients previoucly treated with radiotherapy of head and neck
5. Antifungal or antiviral therapy for oral pathological conditions in the last
6. Other serious concomitant disease
7. History of insulin-dependent Diabetes Mellituss
8. History of oral ulceration, herpes simplex, oral candidiasis, severe gingivitis, active or chronic mucositis or Xerostomia
9. Patients with body weigh >35 kg
10. Women of childbearing potential who are pregnant, breast-feeding or intend to become pregnant
11. Patients with Hepatitis B / C
12. Patients with symptomatic untreated dental infection
13. Patients with oral mucositis grade NCICTC 3 or 4
14. Histological and pathological diagnosis unavailable
15. Patients with signs and symptoms of systemic infection
16. Patient's refusal to sign the informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2012-11; Primary Completion 2014-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
incidence of grade III/IV mucositis | 2 months
  Evaluation of the grade III and IV mucositis incidence in patients undergoing chemo-radiotherapy and taking CD#2 or standard therapy (bicarbonate sodium mouthwash)

SECONDARY OUTCOMES:
percentage of patients able to complete the chemo-radiotherapy treatment | 2 months

OTHER OUTCOMES:
percentage of patients who need enteral nutrition | 2 months from enrolment

CONTACTS AND LOCATIONS:
Overall Officials: Vitaliana De Sanctis, PhD, Principal Investigator — Sant'Andrea Hospital - Radiotherapy Unit
Locations (1):
- Sant'Andrea Hospital, Rome, Rome, Italy